CLINICAL TRIAL: NCT02633995
Title: Spinal Anesthesia in Severe Preeclampsia and Its Impact on Hemodynamics (Case Control Study)
Brief Title: Spinal Anaesthesia and Severe Preeclampsia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, ahmed elsakka, lecturer of anaesthesia faculty of medicine cairo university, Cairo University
Other Study IDs: Mina
Record Dates: First submitted 2015-12-06; First posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- preeclampsia: spinal anaesthesia will be given for cesarean section
  Interventions: Procedure: spinal anaesthesia
- normotensive: spinal anaesthesia will be given for cesarean section
  Interventions: Procedure: spinal anaesthesia

INTERVENTIONS:
Procedure: spinal anaesthesia — regional anesthesia will be induced with a total of 10 mg of 0.5% hyperbaric bupivacaine and 25 µg fentanyl (total volume 2.5 ml) at the L3-4 interspace in the sitting position then the patient will be returned immediately to the supine position with left lateral tilt.

SUMMARY:
The use of spinal anesthesia in pre-eclamptic pregnant woman is of considerable benefit, as these patients present particular hazards with general anaesthesia, such as concerns for rapid airway control and cerebral blood flow alterations during induction of general anaesthesia and intubation However, the incidence of hypotension is high during spinal anesthesia for Cesarean section and it may approach values up to 95 %.

DETAILED DESCRIPTION:
The parturient will be allocated into one of two equal groups (n=30), a severe preeclampsia group (A) and a normotensive group (B). All will receive colload (500 ml voluven) as a coload via wide bore (16 Gauge ) cannula within 5-10 minutes during induction of spinal anesthesia. Standard monitoring with electrocardiography, automated non-invasive arterial pressure (NIAP) measurement, and pulse oximetry will be performed. Systolic arterial pressure (SAP), mean arterial pressure (MAP) and diastolic arterial pressure (DAP) will be monitored. Baseline values will be recorded in the supine position. Central venous line will be inserted in severe preeclampsia group and central venous pressure will be measured every 10 minutes.

Spinal anesthesia will be induced with a total of 10 mg of 0.5% hyperbaric bupivacaine and 25 µg fentanyl (total volume 2.5 ml) at the L3-4 interspace in the sitting position then the patient will be returned immediately to the supine position with left lateral tilt.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 40 years
* Severely Pre-eclamptic females, severe pre-eclampsia is defined as hypertension( BP > 159/109) ,proteinuria ( urinary protein excretion of greater than 5 gm per day) and oliguria(<500 ml in 24 hours) with at least one maternal organ dysfunction .

Exclusion Criteria:

* Age : <18 years
* Obese patients with BMI > 35 Kg/m2
* Preterm delivery
* Patients with contraindication to spinal anesthesia.
* Patients in active labor

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: two equal groups (n=30), Pregnant females with severe pre-eclampsia : (group A) and normotensive parturients (group B) presenting for full term delivery with caesarean section using spinal anesthesia at Kasr Al Aini hospital in the duration of 3 months from december 2015 to march 2016 will be included.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants showing significant hemodynamic changes in response to spinal anesthesia as detected by hemodynamic monitors (blood pressure, heart rate and oxygen saturation) | 3 months

SECONDARY OUTCOMES:
Percentage of participants showing short term adverse side effects in response to spinal anesthesia as nausea, vomiting and shivering | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: maher fawzy, m.d., Study Director — department of anaesthesia faculty of medicine cairo university; nisreen refaie, m.d., Study Chair — department of anaesthesia faculty of medicine cairo university; ahmed elsakka, m.d., Study Chair — department of anaesthesia faculty of medicine cairo university; mina helmy, Principal Investigator — department of anaesthesia faculty of medicine cairo university
Locations (1):
- Cairo University, Cairo, Egypt